CLINICAL TRIAL: NCT02344342
Title: Michigan Advanced Heart Failure TelemoNItoring and FLexible Diuretic Trial - MANIFOLD-HF
Brief Title: University of Michigan Advanced Heart Failure Tele-Monitoring and Flexible Diuretic Project
Acronym: Manifold-HF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The industry sponsor has discontinued the product under evaluation in the study.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Todd M Koelling, MD, Professor of Internal Medicine, Director of Heart Failure Program, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: HUM00091053
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Results first posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-03

CONDITIONS: Heart Failure
Keywords: telemonitoring
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Health Buddy Web Management system (Experimental): Patients randomized to the telemonitoring intervention will be assigned to use the Bosch Health Buddy Web management system.
  Interventions: Device: Telemonitoring; Other: Flexible Diuretic Regimen
- Flexible Diuretic Regimen (Experimental): Patients randomized into the Flexible Diuretic Regimen intervention will have a diuretic regimen specified by specific weight ranges.
  Interventions: Device: Telemonitoring; Other: Flexible Diuretic Regimen

INTERVENTIONS:
Device: Telemonitoring — The Health Buddy web management system allows the patient to enter self-care data through a study provided tablet computer.
  Other Names: Bosch Health Buddy Web Management System
Other: Flexible Diuretic Regimen — Patients will have a prescribed diuretic regimen specified by specific weight ranges.

SUMMARY:
The proposed project is a 2x2 factorial designed study aimed at assessing the impact of 1) a home tele-monitoring system and 2) a flexible diuretic regimen among high risk heart failure patients in the University of Michigan Health System (UMHS).

DETAILED DESCRIPTION:
The proposed project is a 2x2 factorial designed study aimed at assessing the impact of 1) a home tele-monitoring system and 2) a flexible diuretic regimen among high risk heart failure patients in the University of Michigan Health System (UMHS). The first intervention consists of the use of a home monitoring tool utilizing a tablet interface. The device facilitates collection of heart failure patient self-care information, including weight, blood pressure, heart rate and heart failure symptoms. This information is collected and stored on a secured server provided by the vendor, and can be viewed by the physician and nursing team. The second intervention is a flexible diuretic regimen strategy. This intervention will be applied in an independent randomized fashion. The flexible regimen will be prescribed by the patient's physician. The two interventions will be applied to heart failure patients treated at the University of Michigan. A total of 400 patients will be enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

1. University of Michigan patients hospitalized for the treatment of heart failure, within the past 30 days.
2. Patients must be receiving an oral loop diuretic on their home regimen or have received intravenous loop diuretic during the index hospitalization at the time of enrollment.
3. Patients must have an assessment of left ventricular function within the previous 2 years.
4. Patients must have LVEF ≤ 40%, or LVEF >40 with evidence of left atrial enlargement (LA dimension > 40 mm), BNP > 200 ng/ml or PCW > 18 mmHg.

Exclusion Criteria:

* Prisoners
* Residents of long term nursing facilities
* Enrollment into a hospice program
* Receiving dialysis
* Patients with dementia
* Patients with dGFR less than 20ml/min.
* Patients being worked up for heart surgery.
* Patients being worked up for heart transplant.
* Patients being evaluated for revascularization.
* Patients being evaluated for heart valve intervention.
* Patients with primary pulmonary hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-02; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd M Koelling, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized to one of 4 study groups:
  Telemedicine intervention_YES and Flexible Diuretic_YES Telemedicine intervention_YES and Flexible Diuretic_NO Telemedicine intervention_NO and Flexible Diuretic_YES Telemedicine intervention_NO and Flexible Diuretic_NO
Groups:
- Health Buddy Yes and Flexible Diuretic Yes: Telemonitoring: The Health Buddy web management system allows the patient to enter self-care data through a study provided tablet computer.
  Flexible Diuretic Regimen: Patients will have a prescribed diuretic regimen specified by specific weight ranges.
- Health Buddy Yes and Flexible Diuretic Regimen No: Telemonitoring: The Health Buddy web management system allows the patient to enter self-care data through a study provided tablet computer.
  Flexible Diuretic Regimen: These patients will not be assigned to receive a flexible diuretic prescription
- Health Buddy No and Flexible Diuretic Yes: Telemonitoring: These patients will not receive care with the Health Buddy Web intervention.
  Flexible Diuretic Regimen: Patients will have a prescribed diuretic regimen specified by specific weight ranges.
- Health Buddy No and Flexible Diuretic No: Telemonitoring: These patients will not be assigned to the Health Buddy Web intervention.
  Flexible Diuretic Regimen: These patients will not be assigned to follow a flexible diuretic regimen.
Period: Overall Study
Arm/Group | Health Buddy Yes and Flexible Diuretic Yes | Health Buddy Yes and Flexible Diuretic Regimen No | Health Buddy No and Flexible Diuretic Yes | Health Buddy No and Flexible Diuretic No
Started | 13 | 11 | 14 | 13
Completed | 2 | 2 | 0 | 3
Not Completed | 11 | 9 | 14 | 10
Not completed — Industry partner dropped out | 11 | 9 | 14 | 10

BASELINE CHARACTERISTICS:
Population: Group Number of subjects TM_YES_AND_FD_YES 13 TM_YES_AND_FD_NO 11 TM_NO_AND_FD_YES 14 TM_NO_AND_FD_NO 13
Groups:
- Health Buddy Yes and Flexible Diuretic Yes: Telemonitoring: Yes
  Flexible Diuretic Yes
- Health Buddy Yes and Flexible Diuretic No: Telemonitoring: Yes
  Flexible Diuretic No
- Health Buddy No and Flexible Diuretic Yes: Telemonitoring: No
  Flexible Diuretic Yes
- Health Buddy No and Flexible Diuretic No: Telemonitoring: No
  Flexible Diuretic No
- Total: Total of all reporting groups
Arm/Group | Health Buddy Yes and Flexible Diuretic Yes | Health Buddy Yes and Flexible Diuretic No | Health Buddy No and Flexible Diuretic Yes | Health Buddy No and Flexible Diuretic No | Total
Number analyzed (Participants) | 13 | 11 | 14 | 13 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 10 | 8 | 36
  >=65 years | 3 | 3 | 4 | 5 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 5 | 3 | 14
  Male | 9 | 9 | 9 | 10 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 3 | 2 | 3 | 13
  White | 7 | 8 | 11 | 10 | 36
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Hospitalized or Dead in the 180 Day Follow up Period
Description: This is the total combined number of days that all participants in each arm were hospitalized or dead between day 1 and day 180. It is a method to combine the endpoints of death and hospitalization used in heart failure trials. Days hospitalized for all participants are added to days dead for all participants, per arm.
Time Frame: 180 days (6 months)
Population: The subjects included in this measure each completed the 180 follow up period or died within the 180 follow up period. Subjects that had less than 180 days of follow up at the time of study closure are excluded from this analysis.
Measure: Number; unit: Days
Arm/Group | Health Buddy Yes and Flexible Diuretic Yes | Health Buddy Yes and Flexible Diuretic No | Health Buddy No and Flexible Diuretic Yes | Health Buddy No and Flexible Diuretic No
Number analyzed (Participants) | 2 | 2 | 0 | 3
Days | 5 | 23 |  | 0

2. Secondary Outcome: Self Care for Heart Failure Index Score
Description: The self care for heart failure index score ranges from 22 to 88 where 22 is the lowest score meaning cares for oneself least well and 88 means one is most confident or able to care for oneself properly.
Time Frame: 180 day follow up
Population: Two participants completed the study but did not answer all of the questions on this questionnaire, and therefore they are not included in the report for this secondary end point. The subjects included completed the 180 follow up period. Subjects that had less than 180 days of follow up at the time of study closure are excluded from this analysis.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Health Buddy Yes and Flexible Diuretic Yes | Health Buddy Yes and Flexible Diuretic No | Health Buddy No and Flexible Diuretic Yes | Health Buddy No and Flexible Diuretic No
Number analyzed (Participants) | 1 | 2 | 0 | 2
units on a scale | 83 [NA to NA] — For a single participant, there is no range beyond the value of that individual. | 71 [59 to 84] |  | 80 [78 to 81]

3. Secondary Outcome: Minnesota Living With Heart Failure Questionnaire
Description: It provides a total score (range 0-105, where 0 is best quality of life up to 105 as worst Health Related Quality of Life),
Time Frame: 180 day follow up
Population: 2 patients completed the study, whose answers were not coded into the analysis for the questionnaire, therefore they are not included in the report for this secondary end point. The subjects included completed the 180 follow up period. Subjects that had less than 180 days of follow up at the time of study closure are excluded from this analysis.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Health Buddy Yes and Flexible Diuretic Yes | Health Buddy Yes and Flexible Diuretic No | Health Buddy No and Flexible Diuretic Yes | Health Buddy No and Flexible Diuretic No
Number analyzed (Participants) | 1 | 2 | 0 | 2
units on a scale | 49 [NA to NA] — Because there is only a single participant's data presented, there is no range beyond that individual's data. | 22 [15 to 29] |  | 74 [62 to 87]

4. Secondary Outcome: Days to Hospitalization or Death (if it Occurs Within 180 Days)
Description: Time to Hospitalization (if participant was hospitalized and did not die) or death whichever came first. In fact all participants who died in the follow up period were hospitalized first, so actual data reported below also represents time to hospitalization for all participants.
Time Frame: 180 days
Population: All participants who completed 180 days or died prior to 180 days (all who completed study and all listed in all cause mortality)
Measure: Mean (95% Confidence Interval); unit: days till hospitalization
Arm/Group | Health Buddy Yes and Flexible Diuretic Yes | Health Buddy Yes and Flexible Diuretic Regimen No | Health Buddy No and Flexible Diuretic Yes | Health Buddy No and Flexible Diuretic No
Number analyzed (Participants) | 3 | 3 | 2 | 4
days till hospitalization | 107 [62 to 152] | 155 [114 to 195] | 102 [70 to 134] | 122 [83 to 161]

ADVERSE EVENTS:
Time Frame: 180 days (or 6 months) from discharge date or from the day patient started using the intervention.
Description: Subjects were expected to start the intervention on the day of discharge from the hospital, but some subjects once they returned home.
Groups:
- Health Buddy Web YES/Flexible Diuretic YES: Telemonitoring: The Health Buddy web management system allows the patient to enter self-care data through a study provided tablet computer.
  Flexible Diuretic Regimen: Patients will have a prescribed diuretic regimen specified by specific weight ranges.
- Health Buddy Web YES /Flexible Diuretic NO: Telemonitoring: The Health Buddy web management system allows the patient to enter self-care data through a study provided tablet computer.
  Flexible Diuretic Regimen: These patients will not be assigned to receive a flexible diuretic prescription
- Health Buddy Web NO/Flexible Diuretic YES: Telemonitoring: These patients will not receive care with the Health Buddy Web intervention.
  Flexible Diuretic Regimen: Patients will have a prescribed diuretic regimen specified by specific weight ranges.
- Health Buddy Web NO /Flexible Diuretic NO: Telemonitoring: These patients will not be assigned to the Health Buddy Web intervention.
  Flexible Diuretic Regimen: These patients will not be assigned to follow a flexible diuretic regimen.
Arm/Group | Health Buddy Web YES/Flexible Diuretic YES | Health Buddy Web YES /Flexible Diuretic NO | Health Buddy Web NO/Flexible Diuretic YES | Health Buddy Web NO /Flexible Diuretic NO
All-Cause Mortality (participants affected / at risk) | 1/13 | 1/11 | 2/14 | 1/13
Serious Adverse Events (participants affected / at risk) | 5/13 | 4/11 | 7/14 | 6/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/11 | 0/14 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Health Buddy Web YES/Flexible Diuretic YES (N=13) | Health Buddy Web YES /Flexible Diuretic NO (N=11) | Health Buddy Web NO/Flexible Diuretic YES (N=14) | Health Buddy Web NO /Flexible Diuretic NO (N=13)
Congestive heart failure, (Cardiac disorders) | 1 | 0 | 1 | 0 — causing death
Occipital stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — causing death
Hospitalization (Cardiac disorders) | 4 (4) | 3 (3) | 5 (5) | 5 (5) — Heart failure
ventricular tachycardia/ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 — causing death
Death (Cardiac disorders) | 0 | 0 | 1 | 0 — cause unknown

LIMITATIONS AND CAVEATS:
Early termination leading to a small number of subjects analyzed. We have enrolled a total of 51 patients when our target was to enroll 400 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No